CLINICAL TRIAL: NCT05989802
Title: Rapid Research in Diagnostics Development for Tuberculosis Network (R2D2 Kids) and Assessing Diagnostics At Point-of-care for Tuberculosis in Children (ADAPT for Kids)
Brief Title: Rapid Research in Diagnostics Development for TB Network (R2D2 Kids) and Assessing Diagnostics At POC for TB in Children (ADAPT for Kids)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Instituto Nacional de Saúde, Mozambique (Other Government); National Referral Hospital (Other Government); University of Cape Town (Other); Johns Hopkins University (Other); Elizabeth Glaser Pediatric AIDS Foundation (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH); University of California, Irvine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: R01HL169449 (NIH); U01AI152087 (NIH); 7200AA22RFA00004 (Other Grant/Funding Number: USAID)
Record Dates: First submitted 2023-07-28; First posted 2023-08-14 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Tuberculosis; Diagnostics; Global Health
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Evaluation of various novel TB triage and diagnostic tests (Experimental): The investigators will conduct evaluation of novel TB triage and diagnostic tests in a cohort of children with presumed TB. The investigators aim to enroll 250 participants per year at each of three enrollment sites for evaluation of various novel TB triage and diagnostic tests and 30 health workers to assess test usability. Novel test evaluations will be conducted on a rolling basis as new tests ready for field evaluation are identified.
  Interventions: Diagnostic Test: Oral swab molecular testing; Diagnostic Test: Automated Cough Sound Analysis; Diagnostic Test: Automated Lung Sound Analysis; Other: Chest X Ray Computer Aided Detection

INTERVENTIONS:
Diagnostic Test: Oral swab molecular testing — Swab-based testing provides a non-invasive approach to collect respiratory specimens for TB testing. Data in adults suggests that swab-based testing could be valuable when sputum collection is not feasible or available.
Diagnostic Test: Automated Cough Sound Analysis — Cough sounds can be collected through a mobile phone and tablet, and then analyzed with machine learning algorithms to predict TB.
Diagnostic Test: Automated Lung Sound Analysis — Lung sounds can be collected with a non-invasive digital stethoscope, and then saved on a tablet or phone and analyzed by machine learning algorithms to predict TB.
Other: Chest X Ray Computer Aided Detection — Several artificial intelligence algorithms have been developed to predict TB, though this has not yet been validated in children.
  Other Names: Artificial Intelligence algorithm

SUMMARY:
Every year there are an estimated 230,000 childhood deaths from TB. There is an urgent need for novel tests for TB diagnosis in children under 15 years. The Rapid Research in Diagnostics Development for TB Network (R2D2 Kids) and the Assessing Diagnostics at Point-of-care for Tuberculosis in children (ADAPT for Kids) studies seek to reduce the burden of TB worldwide by evaluating faster, simpler, and less expensive TB triage and diagnostic tests for use in children.

DETAILED DESCRIPTION:
The Rapid Research in Diagnostics Development for TB Network (R2D2 Kids) and the Assessing Diagnostics at Point-of-care for Tuberculosis in children (ADAPT for Kids) studies will rigorously assess promising, point-of-care (POC) TB diagnostic tests in clinical studies conducted among children at settings of intended use. There is an urgent need for novel tests for TB diagnosis in children under 15 years because of the challenge of obtaining sputum samples from children and the low sputum bacillary burden among children with TB even when a sample is obtained. This creates delays in diagnosis and treatment initiation, and is a major contributor to the 230,000 childhood deaths from TB each year. Therefore, a non-sputum biomarker-based test has been ranked among the highest priority target product profiles for new TB diagnostics. If inexpensive and simple to perform, such a diagnostic tool could have significant impact by facilitating rapid diagnosis and TB treatment in children. The studies will evaluate the sensitivity and specificity of novel diagnostic tests in children in reference to NIH consensus definitions for childhood TB. In addition, the usability and acceptability of the novel TB diagnostic tests will be assessed through direct observations and surveys of routine health workers.

ELIGIBILITY:
Participant eligibility criteria:

Participants will include children (age <15 years) who present to care with:

A. 2 or more of the following:

* Unexplained cough for any duration
* TB contact or tuberculin skin test or interferon gamma release assay positive
* Abnormal chest X-ray (any abnormality) OR

B. Any one of criteria A AND any one of the following:

* Unexplained weight loss OR unexplained failure to thrive OR Severe Acute Malnutrition
* Unexplained fever ≥2 weeks
* Unexplained lethargy or reduced playfulness ≥2 weeks

The study will exclude participants who:

1. Completed preventive or active TB treatment within the past 12 months (to increase TB prevalence and reduce false-positive results, respectively);
2. Have taken any medication with anti-mycobacterial activity for any reason for greater than 3 days at the time of enrollment (to reduce false-negatives);
3. Are unable to return for follow-up visits; or
4. Whose parents/guardians are unwilling to provide informed consent or who are unwilling to provide assent if applicable (age determined by local IRB)

Assessment of the usability of novel TB tests:

The study will also include health workers at each clinical site who are 1) aged ≥18 years and 2) involved in routine TB testing (collecting specimens for or performing TB tests). Personnel who are unwilling to provide informed consent will be excluded.

Max Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2100 (Estimated)
Dates: Start 2024-01-26 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Proportion with positive index test result among participants with tuberculosis (TB) | 2 years
  Sensitivity - Number with positive index test result/(Number with positive or negative index t test result) among participants with TB. TB will be defined based on a microbiological reference standard (sputum mycobacterial culture results)
Proportion with negative index test result among participants without tuberculosis (TB) | 2 years
  Specificity - Number with negative index test results/(Number with positive or negative index t test result) among participants without TB. TB will be defined based on a microbiological reference standard (sputum mycobacterial culture results)

CONTACTS AND LOCATIONS:
Overall Officials: Adithya Cattamanchi, MD, MAS, Principal Investigator — University of California, Irvine; Nilesh Bhatt, Principal Investigator — Elizabeth Glazer Pediatric AIDS Foundation
Locations (3):
- Instituto Nacional de Saúde, Maputo, Mozambique
- Dora Nginza Hospital, Cape Town, South Africa
- Mulago National Referral Hospital, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Perez-Velez CM, Marais BJ. Tuberculosis in children. N Engl J Med. 2012 Jul 26;367(4):348-61. doi: 10.1056/NEJMra1008049. No abstract available. PMID 22830465
- [Background] World Health Organization. Roadmap towards ending TB in children and adolescents. Geneva: World Health Organization, 2018. Available at: https://www.who.int/tb/publications/2018/tb-childhoodroadmap/en/. Last accessed 1 June 2022.
- [Background] WHO. High-priority target product profiles for new tuberculosis diagnostics: Report of a consensus meeting. Geneva, Switzerland. Available at: http://www.who.int/tb/publications/tpp_report/en/, 2014.
- [Background] Graham SM, Cuevas LE, Jean-Philippe P, Browning R, Casenghi M, Detjen AK, Gnanashanmugam D, Hesseling AC, Kampmann B, Mandalakas A, Marais BJ, Schito M, Spiegel HM, Starke JR, Worrell C, Zar HJ. Clinical Case Definitions for Classification of Intrathoracic Tuberculosis in Children: An Update. Clin Infect Dis. 2015 Oct 15;61Suppl 3(Suppl 3):S179-87. doi: 10.1093/cid/civ581. PMID 26409281
- [Background] World Health Organization. Global Tuberculosis Report 2021. Geneva: World Health Organization, 2021.
- [Background] World Health Organization. Roadmap towards ending TB in children and adolescents. Geneva: World Health Organization, 2018.
- [Background] Lewinsohn DM, Leonard MK, LoBue PA, Cohn DL, Daley CL, Desmond E, Keane J, Lewinsohn DA, Loeffler AM, Mazurek GH, O'Brien RJ, Pai M, Richeldi L, Salfinger M, Shinnick TM, Sterling TR, Warshauer DM, Woods GL. Official American Thoracic Society/Infectious Diseases Society of America/Centers for Disease Control and Prevention Clinical Practice Guidelines: Diagnosis of Tuberculosis in Adults and Children. Clin Infect Dis. 2017 Jan 15;64(2):111-115. doi: 10.1093/cid/ciw778. PMID 28052967
- [Background] WHO consolidated guidelines on tuberculosis: Module 5: Management of tuberculosis in children and adolescents [Internet]. Geneva: World Health Organization; 2022. Available from http://www.ncbi.nlm.nih.gov/books/NBK579387/ PMID 35404556
- [Background] Jaganath D, Beaudry J, Salazar-Austin N. Tuberculosis in Children. Infect Dis Clin North Am. 2022 Mar;36(1):49-71. doi: 10.1016/j.idc.2021.11.008. PMID 35168714
- [Background] Zawedde-Muyanja S, Reuter A, Tovar MA, Hussain H, Loando Mboyo A, Detjen AK, Yuen CM. Provision of Decentralized TB Care Services: A Detect-Treat-Prevent Strategy for Children and Adolescents Affected by TB. Pathogens. 2021 Dec 1;10(12):1568. doi: 10.3390/pathogens10121568. PMID 34959523
- [Background] Dodd PJ, Yuen CM, Sismanidis C, Seddon JA, Jenkins HE. The global burden of tuberculosis mortality in children: a mathematical modelling study. Lancet Glob Health. 2017 Sep;5(9):e898-e906. doi: 10.1016/S2214-109X(17)30289-9. PMID 28807188
- [Background] World Health Organization. High-priority target product profiles for new tuberculosis diagnostics: report of a consensus meeting. Available at: http://apps.who.int/iris/bitstream/handle/10665/135617/WHO_HTM_TB_2014.18_eng.pdf?sequence=12014.
- [Background] Andama A, Whitman GR, Crowder R, Reza TF, Jaganath D, Mulondo J, Nalugwa TK, Semitala FC, Worodria W, Cook C, Wood RC, Weigel KM, Olson AM, Lohmiller Shaw J, Kato-Maeda M, Denkinger CM, Nahid P, Cangelosi GA, Cattamanchi A. Accuracy of Tongue Swab Testing Using Xpert MTB-RIF Ultra for Tuberculosis Diagnosis. J Clin Microbiol. 2022 Jul 20;60(7):e0042122. doi: 10.1128/jcm.00421-22. Epub 2022 Jun 27. PMID 35758702
- [Background] Nkereuwem E, Togun T, Gomez MP, Szekely R, Mace A, Jobe D, Schumacher SG, Kampmann B, Denkinger CM; Reach4KidsAfrica (R4KA) Consortium. Comparing accuracy of lipoarabinomannan urine tests for diagnosis of pulmonary tuberculosis in children from four African countries: a cross-sectional study. Lancet Infect Dis. 2021 Mar;21(3):376-384. doi: 10.1016/S1473-3099(20)30598-3. Epub 2020 Dec 11. PMID 33316214
- [Background] Yellapu GD, Rudraraju G, Sripada NR, Mamidgi B, Jalukuru C, Firmal P, Yechuri V, Varanasi S, Peddireddi VS, Bhimarasetty DM, Kanisetti S, Joshi N, Mohapatra P, Pamarthi K. Development and clinical validation of Swaasa AI platform for screening and prioritization of pulmonary TB. Sci Rep. 2023 Mar 23;13(1):4740. doi: 10.1038/s41598-023-31772-9. PMID 36959347
- [Background] Kevat A, Kalirajah A, Roseby R. Artificial intelligence accuracy in detecting pathological breath sounds in children using digital stethoscopes. Respir Res. 2020 Sep 29;21(1):253. doi: 10.1186/s12931-020-01523-9. PMID 32993620
- [Background] Harris M, Qi A, Jeagal L, Torabi N, Menzies D, Korobitsyn A, Pai M, Nathavitharana RR, Ahmad Khan F. A systematic review of the diagnostic accuracy of artificial intelligence-based computer programs to analyze chest x-rays for pulmonary tuberculosis. PLoS One. 2019 Sep 3;14(9):e0221339. doi: 10.1371/journal.pone.0221339. eCollection 2019. PMID 31479448
- [Background] UCSF Human Research Protection Program. The Level of Review and Minimal Risk. Available at: https://irb.ucsf.edu/levels-review#Category-2-Blood-sampling-limited-amounts. Last accessed 4 Jan 2023.
- [Background] Howie SR. Blood sample volumes in child health research: review of safe limits. Bull World Health Organ. 2011 Jan 1;89(1):46-53. doi: 10.2471/BLT.10.080010. Epub 2010 Sep 10. PMID 21346890